CLINICAL TRIAL: NCT03475420
Title: Compare Patient-centered Outcomes for Lung Cancer Resection Patients Followed With Alternative Intervals of Surveillance Imaging
Brief Title: Post-Treatment Surveillance in Lung Cancer
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: Alliance for Clinical Trials in Oncology (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 17624
Record Dates: First submitted 2018-01-23; First posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- National Cancer Database: Use existing data to define surveillance strategy in use for patients in this cohort. We will use 10 randomly selected lung cancer resection patients from each accredited institution with stage I-III NSCLC (potentially curative resection) diagnosed in 2006-2007 and with 5 years of complete follow up or reported as deceased before 2012.

SUMMARY:
There are 13.7 million Americans currently living with a history of cancer. With continued improvements in cancer treatment and increasing life expectancy, this number is expected to reach nearly 18 million within the next decade. The care of these cancer patients, including surveillance during the post-treatment survivorship phase, is an increasingly important major health care concern and expenditure. As the fourth leading diagnosis among cancer survivors, lung cancer is emerging as a chronic problem that currently affects over 450,000 Americans and is expected to grow by nearly 20% by 2022.

Lung cancer is the second most common cancer in the United States. Of the estimated 182,550 patients newly diagnosed with non-small cell lung cancer (NSCLC) this year, approximately 35% will present with localized disease and be eligible for curative resection. For patients with limited NSCLC, surgical resection is the most effective method of controlling the primary tumor and provides the best opportunity for cure. A recent analysis by this group demonstrated that the number of lung cancer resections has increased over the past decade, with over 45,000 lung cancer resections performed annually in the US.

This research will address a critical gap in knowledge because the optimal approach to post-treatment surveillance following lung cancer resection is unknown. The intensity of recommended surveillance visits ranges from every 3 months during the first two years to an annual visit. Imaging modalities range from CT scans to chest radiographs to no routine imaging for asymptomatic patients. The reason for these significant differences is a lack of quality data on lung cancer surveillance and clinical guidelines based largely on small retrospective analyses and expert opinion.

The National Cancer Data Base (NCDB) provides real world national lung cancer resection and surveillance data on over 70% of newly diagnosed lung cancers from more than 1,500 institutions. This study will compare the effectiveness of the three most common surveillance intensities (CT scans every 3 months vs. 6 months vs. annually) on the stakeholder selected outcome of survival. All analyses will be risk adjusted for differences in patient characteristics at baseline, including tumor characteristics, patient age, comorbid disease, and other potential confounders. Analyses will also be adjusted for the competing risk of death.

DETAILED DESCRIPTION:
This study will use a special study of the National Cancer Database to develop a cohort of NSCLC survivors undergoing surveillance. Cox proportional hazards regression and competing risk analyses will compare the effectiveness of the three most common surveillance intensities (3 months vs. 6 months vs. annually) on survival.

There is also a plan to engage cancer survivors to guide the development of our study comparators, outcomes and demonstration of results.

ELIGIBILITY:
Inclusion Criteria:

* Men or Women
* Diagnosis of surgically resected lung cancer
* American Joint Committee On Cancer (AJCC) stages I-III

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with lung cancer and data available in the National Cancer Database
Sampling Method: Non-Probability Sample
Enrollment: 9613 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Time to Death | Subjects with data from 2006-2007 and with 5 years of complete follow-up or reported as deceased before 2012
  Data elements will include type of surveillance intensity (i.e., 3 month, 6 month or annually) and vital status

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Kozower, MD, Principal Investigator — University of Virginia

IPD SHARING:
Plan to Share IPD: No